CLINICAL TRIAL: NCT04819659
Title: Investigation of the Effect of Pharyngeal Packing on Postoperative Gastric Volume in Patients Undergoing Nasal Surgery
Brief Title: The Effect of Pharyngeal Packing on Postoperative Gastric Volume in Patients Undergoing Nasal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Demet Altun, Assoc. Prof. Dr., Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020/1421; E-29624016-050.99-411338 (Other: istanbul Faculty of Medicine Clin Res Ethics Committee)
Record Dates: First submitted 2021-03-24; First posted 2021-03-29 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Anesthesia; Nasal Surgery; Pharyngeal Packing; Gastric Volume; Postoperative Nausea
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Control (No Intervention): Without pharyngeal pack insertion
- Group Pharyngeal packing (Group PP) (Experimental): Pharyngeal pack insertion after endotracheal intubation
  Interventions: Device: Pharyngeal packing

INTERVENTIONS:
Device: Pharyngeal packing — Placing gauze-like material in the nasal cavity to absorb blood or other fluids right after tracheal intubation.
  Arms: Group Pharyngeal packing (Group PP)

SUMMARY:
Pharyngeal packing is a frequently used application to reduce the incidence and severity of postoperative nausea and vomiting (PONV) in patients who undergo nasal surgery. This study aims to research the effects of PP on gastric antral cross-sectional area (ACSA) and hence gastric volume as assessed by ultrasound, therewithal PONV and sore throat were evaluated as secondary outcomes in rhino logic surgeries (Septorhinoplasty, Septoplasty, Functional endoscopic sinus surgery).

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) after nasal surgery (Septorhinoplasty, Septoplasty, Functional endoscopic sinus surgery) is a very common complication (34-60%). Therefore, pharangeal packing was performed to prevent blood ingestion so as to decrease the incidence of PONV and the risk of aspiration. Also, gastric blood is known to be a powerful emetic. Actually, there is not any evidence in the literature reporting the quantitative values of gastric volumes due to blood ingestion. The aim of this study is to research the effect of pharyngeal packing on the perioperative gastric antral cross-sectional area (ACSA) so the gastric volumes.

Measurements were performed by ultrasound with convex probe in right lateral decubitus position, in order to evaluate the effectiveness of pharyngeal packing in patients undergoing nasal surgery, and to show its effects on PONV and sore throat.

ELIGIBILITY:
Inclusion Criteria:

* undergoing elective nasal or paranasal sinus surgery following overnight fasting
* 18-70 years of age
* accepting to join the study
* American Society of Anesthesiologist (ASA) classification system I-III
* Body mass Index (BMI) < 30 kg/m2

Exclusion Criteria:

* ASA classification higher than III
* Age younger than 18 years
* BMI>30 kg/m2
* Preoperative vomiting or antiemetic medication therapy
* Intubation needing more than two laryngoscopy attempts
* Not agreeing to participate in the study
* Coagulation disorders
* Diseases or conditions affecting gastric volume or motility

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-04-14 (Actual)

PRIMARY OUTCOMES:
The crosssectional area (ACSA) (Postoperative) (mm2) (Postoperative) | 10 minutes before extubation
  measurements are done with USG and calculated with this formula CSA = (AP (anterior-posterior) diameter × CC (cranio-caudal) diameter× 3.14) / 4.

SECONDARY OUTCOMES:
Postoperative presence and severity of PONV | at the first, second and 24th hours in PACU and at the ward
  The severity of PONV was assessed according to the four points score: None (0 point), nausea (1 point), nausea with maximum of two vomiting episodes (2 points), more than two vomiting episodes (3 points).
  When PONV with ≥ 2 points metaclopropamid 10 mg was done, and in order to repetition granisetron 3 mg was added.
The severity of sore throat | at the first, second and 24th hours in PACU and at the ward
  No pain (0 point), mild pain (1 point), moderate pain (2 points) and severe pain (3 points). Patients with severe sore throat were given paracetamol.
Blood volume in the suction system | in the perioperative period
  weighing sponge, pad, compress and blood volume in the aspirator

CONTACTS AND LOCATIONS:
Overall Officials: Demet Altun, Assoc. Prof., Principal Investigator — Istanbul University
Locations (1):
- Istanbul University, Department of Anesthesiology, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Temel ME, Totoz T, Erkalp K, Temel GS, Selcan A. A randomized, double-blind study of the ultrasound assessment of the effect of pharyngeal packing on perioperative gastric volume in nasal surgery. BMC Anesthesiol. 2019 Jul 8;19(1):121. doi: 10.1186/s12871-019-0786-7. PMID 31286899
- [Background] Trotti A, Colevas AD, Setser A, Rusch V, Jaques D, Budach V, Langer C, Murphy B, Cumberlin R, Coleman CN, Rubin P. CTCAE v3.0: development of a comprehensive grading system for the adverse effects of cancer treatment. Semin Radiat Oncol. 2003 Jul;13(3):176-81. doi: 10.1016/S1053-4296(03)00031-6. PMID 12903007